CLINICAL TRIAL: NCT03098290
Title: IDOMENEO: Multimethodical and Multistage Registry-based Longitudinal Study Project to Collect Primary Registry Data and Health Insurance Claims Data of Patients Invasively Treated for Peripheral Artery Disease (PAD) in Germany
Brief Title: IDOMENEO - Is Treatment Reality in Vascular Medicine Evidence-based and Follows Guideline Recommendations? A Project for Quality Development Exemplified by Peripheral Arterial Disease (PAD)
Acronym: IDOMENEO
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: GermanVasc (Other); University Heart Center Hamburg (Unknown); BARMER GEK Germany (Unknown); University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Christian-Alexander Behrendt, Assoc. Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: VF1_2016-028; 01VSF16008 (Other Grant/Funding Number: German Federal Joint Committee); 01VSF18035 (Other Grant/Funding Number: German Federal Joint Committee); DRKS00014649 (Other: German Clinical Trials Registry)
Record Dates: First submitted 2017-03-26; First posted 2017-03-31 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Symptomatic Peripheral Arterial Disease; Occlusive Disease of Artery of Lower Extremity; Quality of Life
Keywords: GermanVasc; Peripheral Arterial Disease; IDOMENEO; Routine Data; Registry Data; Data Validity
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Coronary Artery Bypass; Endarterectomy; Tea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intermittent Claudication: Mild to severe claudication
  Interventions: Procedure: Catheter-based endovascular revascularization; Procedure: Bypass-Surgery; Procedure: Endarterectomy
- Ischaemic Rest Pain
  Interventions: Procedure: Catheter-based endovascular revascularization; Procedure: Bypass-Surgery; Procedure: Endarterectomy
- Critical Limb Threatening Ischaemia: Ulcers, Necrosis, Gangrene
  Interventions: Procedure: Catheter-based endovascular revascularization; Procedure: Bypass-Surgery; Procedure: Endarterectomy

INTERVENTIONS:
Procedure: Catheter-based endovascular revascularization — (e.g. PTA-alone, Bare-Metal or Drug-Eluting-Stent, Covered Stent, Atherectomy, Mechanical Thrombectomy, Scoring Ballon, Cutting Ballon)
  Other Names: ER
Procedure: Bypass-Surgery — Venous or alloplastic or comparable Bypass
  Other Names: Bypass
Procedure: Endarterectomy — Endarterectomy, Patchplasty
  Other Names: TEA

SUMMARY:
The prevalence of peripheral arterial disease (PAD) and the proportion of endovascular procedures for treatment are increasing worldwide. For many cases of treatment or procedures no randomized controlled trials (RCT) or results from meta-analyses are so far available. The decision for treatment and selection of procedure is therefore not uncommonly left up to the personal expertise of the physician. The IDOMENEO study represents a multistage multimethodological project for healthcare research and quality assurance in interdisciplinary vascular medicine, which undertakes a comprehensive examination of this topic. Various methods and data sources (even routine data) are linked in a meaningful way. The essential components of the total project are implementation of a register platform (GermanVasc), which conforms to data protection and data security as well as the development of instruments for valid measurement of the quality of life of patients with PAD. The data protection-conform linking of primary data in the register and routine data of the consortium partner BARMER should also enable validation of the data sources.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic peripheral artery disease (intermittent claudication or critical limb ischemia)
* Invasive treatment (open-surgical or endovascular)
* Informed consent was obtained

Exclusion Criteria:

* No informed consent was obtained
* Acute limb ischemia without any chronic symptomatic PAD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic peripheral artery disease (PAD) treated invasively at certified multidisciplinary vascular centres in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 5608 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
All-cause Mortality | 12 Months
  Death from any reason
Lower Extremity Amputation | 12 Months
  Amputation of lower extremity
Amputation-free Survival | 12 Months
  Long-term-survival without any major amputation
Patency of Revascularization | 12 Months
  Patency of treated vessel
Quality of Life (SF12, WIQ) | 12 Months
  Combined questionnaire including 26 questions using QoL-SF12 and Walking Impairment Questionnaire
Ambulation | 12 Months
Myocardial infarction | 12 Months
Stroke or TIA | 12 Months
Stent or Graft Thrombosis | 12 Months
Functional Status | 12 Months
Modified Rutherford Classification | 12 Months
Foot Infection | 12 Months
Tissue Loss | 12 Months
New Revascularization | 12 Months
Major Adverse Cardiovascular Events (MACE, MACCE) | 12 Months
Major Adverse Limb Events (MALE) | 12 Months
Surgical Site Infection | 12 Months
Major Bleeding Complication | 12 Months
Acute kidney injury (AKI) requiring hemodialysis | At time of discharge (in-hospital period)
  As defined by the National Kidney Foundation.
Ankle-Brachial-Index | 12 Months
Occurrence of target vessel dissection | At time of discharge (in-hospital period)
  Any new dissection of the target vessel related to the procedure
Compartment Syndrome | At time of discharge (in-hospital period)
Graft or Device Failure | At time of discharge (in-hospital period)
Distal Embolisation | At time of discharge (in-hospital period)

CONTACTS AND LOCATIONS:
Overall Officials: Christian-Alexander Behrendt, Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (35):
- Germany (35):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz- und Gefäßzentrum Bad Bevensen, Bad Bevensen
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen (UHZ), Bad Krozingen
  - Charité-Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Asklepios Klinik Birkenwerder, Birkenwerder
  - St. Josef Hospital I Katholisches Klinikum der Ruhr-Universität Bochum, Bochum
  - Gemeinschaftskrankenhaus Bonn, Haus St. Petrus, Bonn
  - GFO Kliniken Bonn, Betriebsstätte St. Marien, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Klinikum Darmstadt GmbH, Darmstadt
  - Städtisches Klinikum Dresden Friedrichstadt, Dresden
  - University Medical Center Düsseldorf, Düsseldorf
  - HELIOS Klinikum Erfurt, Erfurt
  - Elisabeth-Krankenhaus Essen, Essen
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen (UHZ), Freiburg im Breisgau
  - Klinikum Fulda, Fulda
  - University Heart Center Hamburg, Hamburg
  - Agaplesion Diakonieklinikum Hamburg, Hamburg
  - SRH-Klinikum-Karlsbad-Langensteinbach, Karlsbach
  - Klinikum Karlsruhe, Karlsruhe
  - Agaplesion Diakonie Kliniken Kassel, Kassel
  - St. Bonifatius Hospital Lingen, Lingen
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Theresienkrankenhaus Mannheim, Mannheim
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Ev. Krankenhaus Mühlheim an der Ruhr, Mühlheim
  - Isarklinikum München, München
  - Klinikum Peine, Peine
  - Imland Kliniken Rendsburg, Rendsburg
  - Klinikum Rheine I Mathias Spital, Rheine
  - Klinikum Stadt Soest, Soest
  - Klinikum Mutterhaus der Borromäerinnen gGmbH (Mitte), Trier

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Behrendt CA, Riess H, Harter M, Kriston L, Federrath H, Marschall U, Debus ES. [Guideline recommendations and quality indicators for invasive treatment of peripheral arterial disease in Germany : The IDOMENEO study for quality improvement and research in vascular medicine]. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2018 Feb;61(2):218-223. doi: 10.1007/s00103-017-2676-9. German. PMID 29230514
- [Background] Behrendt CA, Härter M, Kriston L, Federrath H, Marschall U, Straub C, Debus ES. [IDOMENEO - Does treatment reality in vascular medicine conform to guidelines and treatment?] Gefaesschirurgie. 2017;22(1):41-47.
- [Background] Behrendt CA, Pridohl H, Schaar K, Federrath H, Debus ES. [Clinical registers in the twenty-first century : Balancing act between data protection and feasibility?]. Chirurg. 2017 Nov;88(11):944-949. doi: 10.1007/s00104-017-0542-9. German. PMID 29079875
- [Background] Behrendt CA, Heidemann F, Haustein K, Grundmann RT, Debus ES; PSI Collaborators. Percutaneous endovascular treatment of infrainguinal PAOD: Results of the PSI register study in 74 German vascular centers. Gefasschirurgie. 2017;22(Suppl 1):17-27. doi: 10.1007/s00772-016-0202-2. Epub 2016 Oct 28. PMID 28715513
- [Background] Behrendt CA, Bertges D, Eldrup N, Beck AW, Mani K, Venermo M, Szeberin Z, Menyhei G, Thomson I, Heller G, Wigger P, Danielsson G, Galzerano G, Lopez C, Altreuther M, Sigvant B, Riess HC, Sedrakyan A, Beiles B, Bjorck M, Boyle JR, Debus ES, Cronenwett J. International Consortium of Vascular Registries Consensus Recommendations for Peripheral Revascularisation Registry Data Collection. Eur J Vasc Endovasc Surg. 2018 Aug;56(2):217-237. doi: 10.1016/j.ejvs.2018.04.006. Epub 2018 May 30. PMID 29776646
- [Background] Riess HC, Debus ES, Schwaneberg T, Hischke S, Maier J, Bublitz M, Kriston L, Harter M, Marschall U, Zeller T, Schellong SM, Behrendt CA. Indicators of outcome quality in peripheral arterial disease revascularisations - a Delphi expert consensus. Vasa. 2018 Oct;47(6):491-497. doi: 10.1024/0301-1526/a000720. Epub 2018 Jun 1. PMID 29856270
- [Background] Behrendt CA, Peters F, Mani K. The Swinging Pendulum of Evidence: Is There a Reality Behind Results from Randomised Trials and Real World Data? Lessons Learned from the Paclitaxel Debate. Eur J Vasc Endovasc Surg. 2020 Apr;59(4):510-511. doi: 10.1016/j.ejvs.2020.01.029. Epub 2020 Feb 20. No abstract available. PMID 32088069
- [Background] Hischke S, Riess HC, Bublitz MK, Kriston L, Schwaneberg T, Harter M, Bertges D, S Debus E, Behrendt CA. Quality Indicators in Peripheral Arterial Occlusive Disease Treatment: A Systematic Review. Eur J Vasc Endovasc Surg. 2019 Nov;58(5):738-745. doi: 10.1016/j.ejvs.2019.06.029. Epub 2019 Sep 13. PMID 31526633
- [Background] Kaschwich M, Behrendt CA, Heydecke G, Bayer A, Debus ES, Seedorf U, Aarabi G. The Association of Periodontitis and Peripheral Arterial Occlusive Disease-A Systematic Review. Int J Mol Sci. 2019 Jun 15;20(12):2936. doi: 10.3390/ijms20122936. PMID 31208079
- [Background] Behrendt CA, Schwaneberg T, Hischke S, Muller T, Petersen T, Marschall U, Debus S, Kriston L. Data Privacy Compliant Validation of Health Insurance Claims Data: the IDOMENEO Approach. Gesundheitswesen. 2020 Mar;82(S 02):S94-S100. doi: 10.1055/a-0883-5098. Epub 2019 May 23. PMID 31121613
- [Background] Behrendt CA, Bjorck M, Schwaneberg T, Debus ES, Cronenwett J, Sigvant B; Acute Limb Ischaemia Collaborators. Editor's Choice - Recommendations for Registry Data Collection for Revascularisations of Acute Limb Ischaemia: A Delphi Consensus from the International Consortium of Vascular Registries. Eur J Vasc Endovasc Surg. 2019 Jun;57(6):816-821. doi: 10.1016/j.ejvs.2019.02.023. Epub 2019 May 22. PMID 31128987
- [Background] Debus ES, Kriston L, Schwaneberg T, Hischke S, Riess HC, Harter M, Marschall U, Federrath H, Behrendt CA. Rationale and methods of the IDOMENEO health outcomes of the peripheral arterial disease revascularisation study in the GermanVasc registry. Vasa. 2018 Oct;47(6):499-505. doi: 10.1024/0301-1526/a000730. Epub 2018 Aug 16. PMID 30113269
- [Result] Aarabi G, Raedel M, Kreutzburg T, Hischke S, Debus ES, Marschall U, Seedorf U, Behrendt CA. Periodontal treatment and peripheral arterial disease severity - a retrospective analysis of health insurance claims data. Vasa. 2020 Mar;49(2):128-132. doi: 10.1024/0301-1526/a000846. Epub 2020 Jan 27. PMID 31983289
- [Result] Behrendt CA, Sedrakyan A, Peters F, Kreutzburg T, Schermerhorn M, Bertges DJ, Larena-Avellaneda A, L'Hoest H, Kolbel T, Debus ES. Editor's Choice - Long Term Survival after Femoropopliteal Artery Revascularisation with Paclitaxel Coated Devices: A Propensity Score Matched Cohort Analysis. Eur J Vasc Endovasc Surg. 2020 Apr;59(4):587-596. doi: 10.1016/j.ejvs.2019.12.034. Epub 2020 Jan 8. PMID 31926836
- [Result] Kreutzburg T, Peters F, Riess HC, Hischke S, Marschall U, Kriston L, L'Hoest H, Sedrakyan A, Debus ES, Behrendt CA. Editor's Choice - Comorbidity Patterns Among Patients with Peripheral Arterial Occlusive Disease in Germany: A Trend Analysis of Health Insurance Claims Data. Eur J Vasc Endovasc Surg. 2020 Jan;59(1):59-66. doi: 10.1016/j.ejvs.2019.08.006. Epub 2019 Nov 16. PMID 31744786
- [Result] Kotov A, Peters F, Debus ES, Zeller T, Heider P, Stavroulakis K, Remig J, Gussmann A, Hoffmann J, Friedrich O, Nolte T, Behrendt CA. The prospective GermanVasc cohort study. Vasa. 2021 Nov;50(6):446-452. doi: 10.1024/0301-1526/a000966. Epub 2021 Jul 19. PMID 34279120
- [Derived] Peters F, Behrendt CA; IDOMENEO Collaborators. Limb Related Outcomes of Endovascular vs. Open Surgical Revascularisation in Patients with Peripheral Arterial Occlusive Disease: A Report from the Prospective GermanVasc Cohort Study. Eur J Vasc Endovasc Surg. 2023 Jul;66(1):85-93. doi: 10.1016/j.ejvs.2023.03.040. Epub 2023 Mar 25. PMID 36972814
- See also: Project website (German) — http://idomeneo.de
- See also: Website of the research group leading the project — http://germanvasc.de